CLINICAL TRIAL: NCT05356611
Title: Engage: A Treatment for Late-Life Depression and Comorbid Executive/Cognitive Dysfunction
Brief Title: Engage for Late-Life Depression and Comorbid Executive Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Brenna Renn, Assistant Professor, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNLV-2022-74
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Depression in Old Age; Psychotherapy; Mild Cognitive Impairment; Executive Dysfunction
Keywords: Older Adults; Late-Life Depression
MeSH Terms: conditions — Cognitive Dysfunction | interventions — engage 8200

STUDY DESIGN:
Intervention Model Description: The trial will be a single-arm feasibility trial of Engage for treatment of late-life depression in older adults with comorbid executive/cognitive dysfunction.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Engage Treatment (Experimental): The study is a single-arm study. The single-arm will be implementation of the 9-week protocol of Engage in an older adult population with late-life depression and comorbid executive dysfunction and mild cognitive impairment.
  Interventions: Behavioral: Engage

INTERVENTIONS:
Behavioral: Engage — Engage is a 9-week, behavioral-based, psychotherapy treatment protocol for late-life depression.

SUMMARY:
Although there are an increasing number of mental health treatment adaptations for older adults, there are still a number of factors to consider when making these adaptations. Cognitive decline is one such factor that places significant burden on older adults and can interfere with traditional mental health therapies. Engage is a behavioral treatment approach that has shown to be effective in treating late life depression. The investigators are testing the feasibility of Engage as a treatment method for late life depression in older adults with cognitive decline. The objective is to corroborate Engage as an alternative late life depression treatment method for a sub-population of older adults with cognitive decline. Cognitive decline poses a unique mental health treatment barrier that is often over looked in younger populations. With a relatively higher prevalence of cognitive decline in older adulthood, it is imperative that a feasible mental health treatment program that can be effective in the presence of cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Ability to read, write, and speak English
* Located in Las Vegas or surrounding area
* Ability to travel to UNLV campus by self or possible caregiver for regular study visits
* Clinically significant symptoms of depression as evidenced by: 1) Scores > 5 on the Geriatric Depression Scale-Short Form (GDS-SF)
* Mild cognitive impairment as evidenced by: 1) Scores > 18 and < 25 on the Montreal Cognitive Assessment (MoCA)

Exclusion Criteria:

* Active suicidal ideation
* History of suicide attempt(s)
* Current symptoms of: 1) Psychosis; 2) Active substance use disorder
* Reported history of: 1) Bipolar disorder ("manic depression"); 2) Intellectual disability
* Currently in or scheduled to initiate individual psychotherapy to avoid treatment interference
* Psychotropic medication permitted if dose was stable over the past 2 weeks
* Currently living in an institutional setting (e.g., assisted living, inpatient, skilled nursing)
* Presence of notable memory-specific cognitive deficits as evidenced by: scores < 9 on the MoCA memory subscale (rendering it difficult to participate in and track/recall events for weekly psychotherapy)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Assessed at Baseline, Week 6, Week 9, and Week 36 follow-up.
  Measure of depressive symptoms used to assess changes across treatment from baseline to mid-treatment, to post-treatment, and follow up at 36 weeks post-baseline. Scores range from 0 - 54 with higher scores indicating worse depression.

SECONDARY OUTCOMES:
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Assessed at Baseline, Week 6, Week 9, and Week 36 follow-up.
  Measure of disability and functioning. Scores range from 0 to 100, with higher scores indicating worse disability.
Behavioral Activation for Depression Scale (BADS) | Assessed at Baseline, Week 6, Week 9, and Week 36 follow-up.
  Measure of behavioral activation (target mechanism). Scores range from 0 to 54, with higher scores indicating more dysfunction.
Social Problem-Solving Inventory Revised-Short Form | Assessed at Baseline, Week 6, Week 9, and Week 36 follow-up.
  measure of problem solving skills. Total scores range from 0 to 100. When all appropriate items are reverse-scored, higher scores indicate better social problem solving functioning.

OTHER OUTCOMES:
Iowa Gambling Task - 2nd Edition | Baseline, Week 9, and Week 36 follow-up.
  Measure of reward response, decision-making and problem solving. Assess changes in target executive functioning skills across treatment. Produces multiple scores, generally with higher scores indicating better decision making.
Hopkins Verbal Learning Memory Test-Revised | Baseline, Week 9, and Week 36 follow-up.
  Measure of memory. Assess potential changes in memory functioning across treatment. Consists of multiple trials and multiple ranges, with higher scores on each trial indicating better memory.
Stroop Color-Word Interference Test | Baseline, Week 9, and Week 36 follow-up.
  Measure of processing speed and response inhibition. Assess changes in target executive functioning skills across treatment. Produces multiple scores across multiple trials and ranges, with higher scores indicating better performance.
Trail Making Test A & B | Baseline, Week 9, and Week 36 follow-up.
  Measure of processing speed and set-shifting. Assess changes in target executive functioning skills across treatment. Time limited task, with higher time indicating worse performance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
The data will be used for the current study. Unidentified data will be available for use within Dr. Brenna Renn's TREATment lab for future lab members to use.